CLINICAL TRIAL: NCT00826306
Title: Comparison of Video-based Versus Written Patient Education on Sunscreen Behavior
Brief Title: Comparison Of Video-based Versus Written Patient Education on Sunscreen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 200816689-1
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Dermatology Disease; Skin Cancer
Keywords: patient education; dermatology patient education; sunscreen; sunscreen education; skin cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video-based education arm (Experimental): Subjects receiving the video-based educational material
  Interventions: Other: Patient Educational Materials
- Written education arm (Active Comparator): Subjects receiving the written educational material
  Interventions: Other: Patient Educational Materials

INTERVENTIONS:
Other: Patient Educational Materials — In the experimental arm, the intervention is the video-based patient educational material on sunscreen. In the active comparison arm (control arm), the comparison intervention is written patient educational material on sunscreen.
  Other Names: Patient educational materials on sunscreen

SUMMARY:
The purpose of this study is to compare the effect of video-based patient education with written instruction on subjects' adherence to sunscreen application.

DETAILED DESCRIPTION:
We plan to conduct a randomized, controlled trial comparing the effect of video-based patient education with written instruction on subjects' adherence to sunscreen application.

Subjects randomized to the video-based education arm will be instructed to watch a video on the importance of sunscreen application and the proper technique of applying sunscreen. Subjects randomized to the written education arm will receive written information on the importance of sunscreen application and the proper technique of applying sunscreen. The contents of the video and the written educational materials will be comparable.

At the end of the study period, 3 months later, subjects will be interviewed via telephone regarding their sunscreen application behavior during the last month of the study period. Subjects will also be interviewed regarding their comprehension and attitude towards video-based and written education materials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent, may be men or women.
* Able to adhere to the study visit schedule and other protocol requirements.
* Capable of giving informed consent.

Exclusion Criteria:

* Non-English speaking individuals
* Individuals with a known allergy to sunscreens
* Individuals with a history of psoriasis, because phototherapy has been shown to be beneficial for their skin condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Sunscreen application behavior. | 3 months

SECONDARY OUTCOMES:
Subjects' comprehension and attitude towards video-based and written education materials. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: April W Armstrong, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Department of Dermatology, Sacramento, California, United States

REFERENCES:
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical/index.html